CLINICAL TRIAL: NCT05140486
Title: Targeted Shortwave Diathermy Combined With Perceptual Training for Patients With Severe Traumatic Optic Neuropathy After Endoscopic Optic Nerve Decompression: a Preliminary Clinical Trial.
Brief Title: Targeted Shortwave Diathermy Combined With Perceptual Training for Patients With Severe Traumatic Optic Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Qingping Tang, Director, Hunan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HunanPPH
Record Dates: First submitted 2021-02-01; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Traumatic Optic Neuropathy
Keywords: Shortwave diathermy; perceptual training; traumatic optic neuropathy
MeSH Terms: conditions — Optic Nerve Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shortwave diathermy and perceptual training (Experimental): The subjects in this group will receive shortwave diathermy 5 days per week for 4 weeks and perceptual training 5 days per week for 10 weeks after endoscopic optic nerve decompression surgery.
  Interventions: Procedure: Rehabilitation: shortwave diathermy and perceptual training
- Nonrehabilitation (No Intervention): The subjects in the nonrehabilitation group will not only receive any rehabilitation therapy after endoscopic optic nerve decompression surgery.

INTERVENTIONS:
Procedure: Rehabilitation: shortwave diathermy and perceptual training — All subjects in the rehabilitation group received shortwave diathermy therapy 5 days per week for 4 weeks and perceptual training 5 days per week for 10 weeks.
  Arms: Shortwave diathermy and perceptual training

SUMMARY:
Purpose: Patients with severe traumatic optic neuropathy (TON) have limited improvement in visual function despite therapy. The hypothesis of the study is that the targeted shortwave diathermy combined with perceptual training may enhance visual function in patients with severe TON after endoscopic optic nerve decompression (EOND) surgery.

Design: Clinical trial Subjects: Twenty-two subjects with severe TON after EOND surgery were randomly assigned to either a rehabilitation (Reh) group or nonrehabilitation (Nreh) group.

Methods: High-resolution computed tomography and MRI were used to locate the impaired nerve. The subjects in the Reh group received targeted shortwave diathermy therapy 5 days per week for 4 weeks and perceptual training 5 days per week for 10 weeks.

Main Outcome Measures: A thorough evaluation of visual function, visual evoked potential, and diffusion tensor imaging was executed.

DETAILED DESCRIPTION:
Study sample description Indirect traumatic optic neuropathy (TON) was diagnosed by a history of blunt head or facial trauma combined with decreased visual acuity, color vision and a relative afferent pupillary defect with a normal fundus during the early period of post-trauma. The investigators excluded cases with direct trauma to optic nerve identified by high-resolution CT scan of the orbital and optic canal. The patients with indirect TON were intravenously administered methylprednisolone (30 mg/kg per day) every day for three consecutive days. All consecutive subjects with indirect TON who were admitted to Xiangya Hospital and managed with endoscopic optic nerve decompression surgery were recruited. The subjects were randomly assigned to either a rehabilitation group or a nonrehabilitation group. Since there were no grading criteria in evaluating the severity of indirect TON, TON with Best-corrected visual acuity equal to or more than 1.85 LogMAR after endoscopic optic nerve decompression surgery was considered severe TON and those patients were recruited in this study. The subjects in the rehabilitation group will receive shortwave diathermy therapy and perceptual training after endoscopic optic nerve decompression surgery. The subjects in the nonrehabilitation group will not receive any rehabilitation treatment after endoscopic optic nerve decompression surgery.

Endoscopic ON decompression surgery All operations were performed under general anesthesia by a surgeon (Hua Zhang). Briefly, a routine endoscopic endonasal sphenoethmoidectomy was performed to expose and resect the posterior ethmoidal lamina papyracea. After the optic canal was exposed, the upper, medial and partial lower surfaces of the whole range of the optic canal wall were removed. Finally, the ON sheath from the annulus of the Zinn to the cranial cavity, along with the annulus of the Zinn, was incised, and the surface of the ON was covered with a piece of gelatin sponge filled with methylprednisolone solution (40 mg/mL).

Shortwave diathermy therapy The Shortwave diathermy (SWD) device applied in this study was DL-CⅡ (Dajia®, Shantou, China). This therapeutic apparatus delivered at a frequency of approximately 27.12±0.6% MHz in continuous modes with a power of 50 W±20%. In our study, two sets of circular capacitive electrodes were used with a diameter of 80 mm for adults and 50 mm for children. The fracture areas were located using high-resolution CT scan. One electrode was applied in the temporal area of the ipsilateral side of the injured nerve identified by a three-dimensional alignment procedure through high-resolution CT scan. This area was not only shorter distance from the skin to the injured nerve but was also as far away from the crystalline lens as possible. To decrease the negative effects of SWD on the nerve systems, another circular electrode of SWD was applied in the frontal area of the ipsilateral side of the injured nerve. In the acute stage of the TON (within 10 days after injury), the athermal mode of the SWD was applied to the marked areas for a 10-minute daily session. Ten days after injury, the microthermal mode was used for a 15-minute daily session. All subjects in the rehabilitation group received SWD therapy 5 days per week for 4 wks.

Perceptual training Perceptive learning sessions were composed of a series of training procedures. First, sensory stimulations including touch, stroking, tapping and pressing on the local area of the ipsilateral eye as well as surface location of the injured ON were offered. Second, light stimulation was applied at different intensities of bright based on evaluation of the pupillary light reflex of the subject, 1 to 5 seconds each time, 10 to 15 times a day, and avoiding glare and longtime light stimulation on eye when training. Additionally, the subjects were instructed to enter the bright room from the dark room when the participants were wearing an eye patch in the intact eye. Third, differentiation of the shapes and objects in dynamic or static states with different colors, different sizes and different shapes was performed. Either real objects or pictures could be selected in the training session. Fourth, different written words with different sizes and different distances were discriminated in the different directions of the eye. Based on evaluation of the visual acuity, the training sequence was from large words to small, from simple words to complex, and from proximal to distal distance of the eye. Fifth, color vision was trained using real objects or pictures. The subjects were instructed to select the color from the single and bright to multiple and dark color. The color contrast was initiated from maximum to minimal contrast. Finally, the visual field training was scattered in the above training methods. Each training media including the light, objects, words and color was input from the anterior, superior, inferior, nasal and temporal sides of the eye. These trainings started from the center of the normal visual field to the terminal of the visual field. When the training media reached the terminal of the visual field in every direction, ocular fixation with 2-5 seconds was performed to increase the scope of the visual field. Each stimulation was given 5-10 times for each direction. In the early periods of the training, when the visual acuity was complete loss, the training sections were relatively independent. When the visual acuity of subjects was partially recovered, the training sections were mixed. In addition, many training techniques were used in this study. First, visual imagery training was used when the patients had complete or severe visual loss. Visual imagery training can be defined as "a dynamic state during which the representation of a specific object is internally reactivated within visual memory without any overt visual input and that is governed by the principles of central visual control". The intervention of the VI training was as follows: the subjects used the intact eye to observe the object for 5 seconds, then the participants closed their eyes and imagined viewing the object using the injured eye for 10 seconds for 10 repetitions. Additionally, proprioceptive training, including going over the barriers, going up and downstairs, walking the slope, and training the balance, was executed. Finally, constraint-induced perceptive therapy was performed when the visual lesion partially recovered. The subjects wore an eye patch on the intact eye for 30 minutes in one section, 2 to 4 hours a day, 7 days per week. In constraint-induced perceptive training, activities of daily living (ADL), natural environmental training and fun games with colorful objects were executed, and the subjects were instructed to complete the ADL, play gobang, watch the green leaves and colorful flowers from proximal to distal distance. All the subjects in the Reh group received perceptive learning therapy 5 days per week for 10 weeks except constraint-induced perceptive therapy.

ELIGIBILITY:
Inclusion criteria:

The indications for endoscopic optic nerve decompression surgery included no improvement after intravenous treatment for 24 hours, no evidence of injury in the intracranial portion of the optic nerve, and the presence of bony fragments or hematoma compressing the optic nerve.

TON with best-corrected visual acuity equal to or more than 1.85 logMAR after surgery was considered as severe TON, and those patients managed with endoscopic optic nerve decompression surgery were recruited in this study.

Eligible criteria for the participants were as follows: (1) not receiving other physical therapy regimens aside from this intervention; (2) age 3 to 60 years old; (3) ability to execute simple verbal instructions; (4) not being delirious; (5) having stable vital signs and medical conditions.

Exclusion criteria:

The exclusion criteria included severe diffuse brain damage, and/or severe cardiac and pulmonary disease, which were contraindicated in rehabilitation procedure.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI | 15 minutes
  A 32-channel head coil on a 3.0T MRI system (Philips, Ltd, Best, the Netherlands) was used for the acquisition of imaging data. T1- and T2-weighted, fat-suppressed images were obtained axially through the orbit and some parts of the brain, including the intracranial portion of the optic nerve, postoperatively and 10 weeks after rehabilitation.
Diffusion tensor imaging | 15 minutes
  Optic nerve diffusion tensor imaging images were obtained using single-shot echoplanar imaging sequences. The images were acquired from the optic papilla to the orbital apex of the optic nerve with 40 contiguous slices. The region of interest was manually manually placed over the optic nerve at the anterior, middle, and posterior segments on the non-diffusion-weighted image. The fraction anisotropy, mean diffusivity, axial diffusivity, and radial diffusivity of optic nerves were measured.

SECONDARY OUTCOMES:
Visual evoked potential | 30 minutes
  Pattern visual evoked potential testing was recorded using an MEB-9404C (Nihon Kohden Corp, Tokyo, Japan). The latency and amplitude of the P100 wave in the VEP testing were collected for analysis.
Best-corrected visual acuity | 5 minutes
  Best-corrected visual acuity was measured by a standardized Snellen visual chart. Visual results were converted into logMAR units for the convenience of statistical analysis. Hand motion, light perception, and no light perception were converted to 2.3, 2.5, and 3 logMAR units, respectively.
Color vision | 5 minutes
  Color vision was evaluated using the Ishihara color vision test 24 plate. The exclusion criterion of the color vision test was congenital color vision deficiency. The number of correct answers in a set of 24 plates was recorded as the color vision score.

CONTACTS AND LOCATIONS:
Overall Officials: XiaoYe Wang, Study Chair — Brain Hospital of Hunan Province, Hunan University of Chinese Medicine
Locations (1):
- Tang, Changsha, China

IPD SHARING:
Plan to Share IPD: No